CLINICAL TRIAL: NCT01224678
Title: Vitamin D and Breast Cancer Biomarkers
Brief Title: Vitamin D and Breast Cancer Biomarkers in Female Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CALGB-70806; CALGB-70806; CDR0000687263 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2010-10-19; First posted 2010-10-20 (Estimated); Results first posted 2018-06-25 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Patients receive oral placebo once daily for 12 months.
  Interventions: Other: placebo
- Vitamin D (Experimental): Patients receive oral vitamin D (2000 IU) once daily for 12 months.
  Interventions: Dietary Supplement: vitamin D

INTERVENTIONS:
Dietary Supplement: vitamin D — Given orally
  Arms: Vitamin D
Other: placebo — Given orally
  Arms: Placebo

SUMMARY:
RATIONALE: Vitamin D may help prevent breast cancer.

PURPOSE: This randomized clinical trial is studying vitamin D and breast cancer biomarkers in female patients.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate change in mammographic density using the Boyd method after one year of vitamin D supplementation compared to placebo in premenopausal women.

Secondary

* To explore changes in the serum biomarker IGF1 in response to one year of vitamin D or placebo supplementation in premenopausal women.
* To explore changes in cellular proliferation (atypia and Ki67) in response to one year of vitamin D or placebo supplementation in premenopausal women.
* To explore correlations between change in breast cancer biomarkers (density, IGF1, atypia, and Ki67) with each other and with change in vitamin D levels.
* To compare methods of mammographic density analysis.
* To validate a recently developed sunlight questionnaire.

OUTLINE: This is a multicenter study. Patients are stratified according to baseline vitamin D (sufficient [≥ 30 ng/mL or ≥ 75 mmol/L] vs insufficient [< 30 ng/mL or < 75 mmol/L]) and institutional random periareolar fine-needle aspiration (RPFNA) status (performs RPFNA vs does not perform RPFNA). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral placebo once daily for 12 months.
* Arm II: Patients receive oral vitamin D (2000 IU) once daily for 12 months. Tissue and blood samples are collected at baseline and at 12 months for laboratory biomarker analysis. Patients also complete questionnaires at baseline and at 12 months.

ELIGIBILITY:
1. Premenopausal women 55 years of age or younger with regular menstrual cycles (at least four cycles in the last six months). Women with fewer than 4 menses in the last 6 months or who have had a hysterectomy with ovaries intact will be considered premenopausal if FSH level < 20.
2. Women with breast density ≥ 25% (scattered fibroglandular densities or greater) are eligible.
3. Prior Treatment

   1. Patients who are currently receiving hormone replacement therapy (estrogen or progesterone); or are taking tamoxifen or raloxifene are not eligible. Women who have taken these medications must have stopped for at least 4 months prior to study entry.

      Topical estrogen (eg, transdermal patches and vaginal estrogens) is allowed.
   2. Patients who are currently using hormonal contraception, should be taking it for at least 4 months prior to study entry.
4. Vitamin D Use

   1. Patients who are taking regular vitamin D supplementation (above 400 IUs daily) and refuse or are unable to stop use are not eligible. Women who agree to stop will need to do so for at least 6 months prior to registration.
   2. Patients may not start vitamin D supplementation after registration (regardless of results of vitamin D testing) but they may continue vitamin D if they are already taking 400 IUs daily or less and have been taking vitamin D for at least 6 months prior to baseline mammogram.
5. Patients with a history of breast cancer (including DCIS) or ovarian cancer are not eligible.
6. Patients with a history of breast implants or breast reduction are not eligible.
7. Patients with two or more bone fractures in the past five years are not eligible.
8. Patients with a diagnosis of osteoporosis with physician recommendation for treatment of low bone mass are not eligible.
9. Patients known to have hyperparathyroid disease or other serious disturbances of calcium metabolism requiring intervention in the past 5 years are not eligible.
10. Patients with a history of kidney stones (unless documented not to have been a calcium stone) are not eligible.
11. Patients participating in a concurrent breast cancer chemoprevention trial are not eligible.
12. Required initial laboratory values - Calcium < 10.5 mg/dL

Max Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie E. Wood, MD, Study Chair — University of Vermont
Locations (103):
- United States (103):
  - Regional Medical Center, Anniston, Alabama
  - Contra Costa Regional Medical Center, Martinez, California
  - Camino Medical Group - Treatment Center, Mountain View, California
  - El Camino Hospital Cancer Center, Mountain View, California
  - Bay Area Breast Surgeons, Incorporated, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee, Incorporated, Oakland, California
  - Palo Alto Medical Foundation, Palo Alto, California
  - Pismo Beach, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - Bendheim Cancer Center at Greenwich Hospital, Greenwich, Connecticut
  - Michael and Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Michiana Hematology-Oncology, PC - Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Michiana Hematology Oncology PC - Plymouth, Plymouth, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC - La Porte, Westville, Indiana
  - National Naval Medical Center, Bethesda, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at South Shore, South Weymouth, Massachusetts
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - New Hampshire Oncology - Hematology, PA at Payson Center for Cancer Care, Concord, New Hampshire
  - New Hampshire Oncology - Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Lakes Region General Hospital, Laconia, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Charles R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - Mount Sinai Medical Center, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Faxton Regional Cancer Center, Utica, New York
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Duke Cancer Institute, Durham, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Rex Cancer Center at Rex Hospital, Raleigh, North Carolina
  - Rex Cancer Center of Wakefield, Raleigh, North Carolina
  - Zimmer Cancer Center at New Hanover Regional Medical Center, Wilmington, North Carolina
  - Forsyth Regional Cancer Center at Forsyth Medical Center, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Cancer Care Associates - Mercy Campus, Oklahoma City, Oklahoma
  - Cancer Centers of the Carolinas - Faris Road, Greenville, South Carolina
  - Greenville Hospital Cancer Center, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Seneca, Seneca, South Carolina
  - Cancer Centers of the Carolinas - Spartanburg, Spartanburg, South Carolina
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Doctor's Hospital of Laredo, Laredo, Texas
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: Yes
Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive
URL: https://nctn-data-archive.nci.nih.gov/

REFERENCES:
- Available data/document: Individual Participant Data Set — https://nctn-data-archive.nci.nih.gov/ — Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Vitamin D
Started | 150 | 150
Completed | 150 | 150
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients were used for baseline analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vitamin D | Total
Number analyzed (Participants) | 150 | 150 | 300
Age, Continuous [Median (Full Range); unit: years] | 44.3 [24.8 to 55.1] | 42.7 [22.7 to 59.4] | 43 [22.7 to 59.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 150 | 300
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 23 | 42
  Not Hispanic or Latino | 129 | 124 | 253
  Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 9 | 5 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 14 | 21 | 35
  White | 124 | 114 | 238
  More than one race | 1 | 4 | 5
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 150 | 150 | 300

OUTCOME MEASURES:

1. Primary Outcome: Percent Change (Between Baseline and Month 12) in Mammographic Density by the Boyd Method Compared Between Arms
Description: To evaluate change in mammographic density using the Boyd method after one year of vitamin D supplementation compared to placebo in premenopausal women. The percent change in breast density will be reported here.
Time Frame: 12 months
Population: 86 of the 300 patients were analyzed for the primary endpoint
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 46 | 40
percent change | -3.4 (7.1) | -1.4 (11.9)

ADVERSE EVENTS:
Arm/Group | Placebo | Vitamin D
Serious Adverse Events (participants affected / at risk) | 0/150 | 0/150
Other Adverse Events (participants affected / at risk) | 1/150 | 1/150
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=150) | Vitamin D (N=150)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (9) | 1 (7)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (20) | 1 (18)
Vomiting (Gastrointestinal disorders) | 1 (7) | 1 (10)
Pain (General disorders) | 0 (0) | 1 (1)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (2) | 0 (0)
GGT increased (Investigations) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (6)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1)
Headache (Nervous system disorders) | 1 (50) | 1 (49)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (2)
Irregular menstruation (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less